CLINICAL TRIAL: NCT02862288
Title: Preliminary Study of Microwave Tumoral Ablation Performances for the Treatment of Pulmonary, Renal and Bone Neoplasia.
Acronym: TherMO
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: API/2011/23
Record Dates: First submitted 2016-08-01; First posted 2016-08-11 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-08

CONDITIONS: Lung Tumor; Bone Tumor; Renal Tumor
MeSH Terms: conditions — Lung Neoplasms; Bone Neoplasms; Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Renal tumor (Experimental): Microwave ablation of renal tumor
  Interventions: Device: Microwave ablation with Acculis Accu2i pMTA Applicator
- Lung tumor (Experimental): Microwave ablation of lung tumor
  Interventions: Device: Microwave ablation with Acculis Accu2i pMTA Applicator
- Bone tumor (Experimental): Microwave ablation of bone tumor
  Interventions: Device: Microwave ablation with Acculis Accu2i pMTA Applicator

INTERVENTIONS:
Device: Microwave ablation with Acculis Accu2i pMTA Applicator

SUMMARY:
The aims of this work were to assess the feasibility, efficacy, short-term outcome and safety of microwave ablation in the treatment of malignant bone, lung and renal tumors.

ELIGIBILITY:
Inclusion Criteria:

* Men and women > 18 years old
* Thermoablation indication of renal neoplasia, bone or lung decided during a multidisciplinary consultation meeting - Generally speaking, the indications are: (i) inoperable primary malignant tumor or secondary malignant tumor, (ii) resectable primary malignant renal and lung tumor with medical contraindication to surgery or general anesthesia
* Signature of informed consent for participation
* Affiliation to a social security scheme or French beneficiary of such a regime.

Exclusion Criteria:

* Contraindication to percutaneous thermoablation
* Renal or lung tumor up to 4 cm
* Women of childbearing age, premenopausal, non-sterilized surgically, and unwilling to use effective contraception
* Legal incapacity or legal capacity limited
* Person unlikely to cooperate in the study and / or low degree of cooperation expected by the investigator
* Person without health insurance
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-09; Primary Completion 2015-02 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Tumor necrosis rate in post-intervention over one month monitoring period. | one month

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien Aubry, M.D., Principal Investigator — Centre hospitalier régional universitaire de Besançon
Locations (1):
- CHU Besançon, Besançon, France

IPD SHARING:
Plan to Share IPD: No